CLINICAL TRIAL: NCT03305601
Title: Information During Maternity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMARTMATER
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: application on smarthphone — application on smarthphone

SUMMARY:
During the pregnancy , it's now compulsary for the doctors to inform pregnant women and the couple about the medical, non medical informations and explain the physiological changes . As usual, medical staff and doctors explain and inform by oral and with a booklet patient.

In order to cluster and make more accessible these informations, the maternity team of GHPSJ has developed an application on smartphone . If this application has been evaluated on his contents and accordance to recommendations, there is no evaluation about the satisfaction of patient.

The aim is to study the impact of this kind of application on pregnant women satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* delivery at 37 weeks of amenhorrhea
* age > 18
* with an email address

Exclusion Criteria:

* refusing participation
* foetal pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 104 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
satisfaction score | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France